CLINICAL TRIAL: NCT04722367
Title: Being Present With Art: The Impact of Mindful Engagement With Art on Awareness and Connection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2000028825
Record Dates: First submitted 2021-01-19; First posted 2021-01-25 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Stress
Keywords: art pedagogy; mindfulness
MeSH Terms: interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Art Pedagogy and Mindfulness (Experimental): Each participant will take part in four 1-hour sessions. Study activities include guided meditation, close looking, drawing, writing, and storytelling. Each session will begin with a guided meditation that is followed by an exercise inspired by two works of art, and end with an opportunity for students to reflect on the experience.
  Interventions: Behavioral: Art Pedagogy and Mindfulness

INTERVENTIONS:
Behavioral: Art Pedagogy and Mindfulness — Each participant will take part in four 1-hour sessions. Study activities include guided meditation, close looking, drawing, writing, and storytelling. Each session will begin with a guided meditation that is followed by an exercise inspired by two works of art, and end with an opportunity for students to reflect on the experience.

SUMMARY:
The purpose of this study is to observe and measure the impact of mindfulness and art pedagogy on stress levels amongst students.

DETAILED DESCRIPTION:
This study uses a waitlist control design. Participants will be randomly assigned to either session one or session two.

Regardless if they are registered for Session One or Session Two, each participant will be invited to self-report their stress levels, feelings of being aware of the present moment, and feelings of connection and belonging on a weekly basis. There will be a follow-up survey at the end of Session One and Session Two to compare changes between participants who have already received the intervention and those who have not. In this way, Session One participants act as a control group. This follow-up survey will be utilized once again after Session Two finishes in order to examine whether there is a lasting impact on Session One participants.

ELIGIBILITY:
Inclusion Criteria:

* Yale student
* 18 years of age or older
* Must complete all survey measures
* Must be available Mondays 5-6 pm EST in October and November

Exclusion Criteria:

* Not a Yale student
* Not 18 years of age or older
* Does not complete all survey measures
* Not available Mondays 5-6 pm EST in October and November

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Change in stress from Impact of Being Present with Art Intervention | Baseline, 4 weeks
  A primary objective of this study is to determine whether mindful engagement with art reduces student stress levels. This will be measured by the Perceived Stress Scale (min = 0; max = 4) which consists of 10 scale items. The higher the score, the more likely participants are stressed. Participants who received the intervention in Session One will be compared to the control (Session Two).
Change in mindfulness from Impact of Being Present with Art Intervention | Baseline, 4 weeks
  A primary objective of this study is to determine whether mindful engagement with art increases mindful awareness in students. This will be measured by the Mindful Awareness Scale (min = 1; max = 6) which includes 15 questions. The higher the score, the more mindful participants are. Participants who received the intervention in Session One will be compared to the control (Session Two).
Change in Connectedness from Impact of Being Present with Art Intervention | Baseline, 4 weeks
  A primary objective of this study is to determine whether mindful engagement with art increases feelings of connectedness in students. This will be measured by a scale created by the investigators to ask participants how connected they feel to the Yale community (min = 1; max = 5). This scale involves one question. The higher the score, the more connected participants feel to the Yale community. Participants who received the intervention in Session One will be compared to the control (Session Two).

SECONDARY OUTCOMES:
Change in Longitudinal Impact of Being Present with Art Intervention on Stress | Baseline, 4 weeks, 8 weeks
  A secondary objective of this study is to determine whether the Being Present with Art intervention resulted in a longitudinal decrease in stress for Session One participants. This outcome is measured by the Perceived Stress Scale (min = 0; max = 4) which consists of 10 scale items. The higher the score, the more stressed participants are.
Change in Longitudinal Impact of Being Present with Art Intervention on Mindfulness | Baseline, 4 weeks, 8 weeks
  A secondary objective of this study is to determine whether the Being Present with Art intervention resulted in a longitudinal increase in mindfulness for Session One participants. This outcome is measured by the Mindful Awareness Scale (min = 1; max = 6) which consists of 15 scale items. The higher the score, the more mindful participants are.
Change in Longitudinal Impact of Being Present with Art Intervention on Connectedness | Baseline, 4 weeks, 8 weeks
  A secondary objective of this study is to determine whether the Being Present with Art intervention resulted in a longitudinal increase in connectedness for Session One participants. This outcome is measured by connectedness scale we created for the purpose of this study (min = 1; max = 5) which consists of one question. Higher scores indicate increased participant feelings of connectedness to the Yale community.

OTHER OUTCOMES:
Pre vs. Post-Session Check-In: Investigating Stress | Session One: Week 1, Week 2, Week 3, Week 4; Session Two: Week 5, Week 6, Week 7, Week 8
  Session One and Session Two participants each attended 4 consecutive weeks of the Being Present with Art programming. The investigators wanted to know whether stress measures before vs. after any one of these four sessions resulted in decreased stress for both Session One and Session Two participants. This was measured by asking students one question about how stressed they currently felt (min = 0; max = 4). Higher scores indicate increased participant stress.
Pre vs. Post-Session Check-In: Investigating Mindfulness | Session One: Week 1, Week 2, Week 3, Week 4; Session Two: Week 5, Week 6, Week 7, Week 8
  Session One and Session Two participants each attended 4 consecutive weeks of the Being Present with Art programming. The investigators wanted to know whether mindfulness measures before vs. after any one of these four sessions resulted in increased mindfulness for both Session One and Session Two participants. This was measured by asking students one question about how aware of the present moment they currently felt (min = 0; max = 4). Higher scores indicate increased mindful awareness.
Pre vs. Post-Session Check-In: Investigating Connectedness | Session One: Week 1, Week 2, Week 3, Week 4; Session Two: Week 5, Week 6, Week 7, Week 8
  Session One and Session Two participants each attended 4 consecutive weeks of the Being Present with Art programming. The investigators wanted to know whether connectedness measures before vs. after any one of these four sessions resulted in increased connectedness for both Session One and Session Two participants. This was measured by asking students one question about how connected to the Yale community they currently felt (min = 0; max = 4). Higher scores indicate increased feelings of connectedness.

CONTACTS AND LOCATIONS:
Overall Officials: Laurie Santos, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States